CLINICAL TRIAL: NCT02084550
Title: Amino Acids in Ileal Pouch-anal Anastomosis for Ulcerative Colitis: a Randomized, Assessor-blinded, Placebo-controlled Trial
Brief Title: Amino Acids in Ileal Pouch-anal Anastomosis for Ulcerative Colitis
Acronym: AMINOPOUCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Anders Mark Christensen, PhD student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1-10-72-48-14
Record Dates: First submitted 2014-03-05; First posted 2014-03-12 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — amino-acid, glucose, and electrolyte solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaminolac (Active Comparator): Intravenous Vaminolac during 3 hours, with an infusion rate of 1,6ml/kilogram bodyweight/h.
  Interventions: Dietary Supplement: Vaminolac
- Saline (Placebo Comparator): Intravenous saline during 3 hours, with an infusion rate of 1,6ml/kilogram bodyweight/h.
  Interventions: Other: Saline

INTERVENTIONS:
Dietary Supplement: Vaminolac — Vaminolac with an amino acid content corresponding humane breast milk.
  Arms: Vaminolac
Other: Saline — Intravenous isotonic saline with a sodium chloride content of 9mg/ml.
  Arms: Saline

SUMMARY:
The detrimental effects of catabolism, insuline resistance and muscle wasting on surgical outcome is wellknown. This catabolism is especially pronounced in patients with acute or chronic inflammation (IBD, cancer) and for those undergoing major surgery. Patients with ulcerative colitis operated with an ileal pouch-anal anastomosis (j-pouch) fall well into both these categories.

To prevent this undesirable catabolism, we will investigate the effects of intravenous administration of predominantly anabolic amino acids (with an amino acid content equal to breast milk) on whole body metabolism, with special emphasis on muscle and fat metabolism and intracellular signalling pathways.

Twenty-four patients will be block-randomized by gender in this parallel-group, randomized, assessor-blinded, placebo-controlled trial to receive either Vaminolac® (Fresenius Kabi) or saline. Metabolism before and after the intervention will be assessed by palmitate- and amino acid kinetics of radioactively labelled tracers, while muscle and fat biopsies will be analyzed for differences in intracellular signaling pathways (PI3 kinase, Akt, etc.) as a measure of cellular activity.

With this study we hope to find evidence for anabolic effects of intravenous amino acids in j-pouch surgery for ulcerative colitis. The perspective is a potential for primary prophylaxis of surgical complications, reduction in the length of hospitalization, and subsequently optimized long-term functional outcome of the pouch.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulcerative colitis who are having an ileal pouch-anal anastomosis performed, 18 < age < 50, written informed consent.

Exclusion Criteria:

* Inability to understand written Danish, postmenopause, severe asthma, diabetes mellitus, severe rheumatologic disease, severe comorbidity (ASA group III-IV) in general. Acute or progressing liver failure, uremia without possibility for dialysis, phenylketonuria, defects in amino acid metabolism. Participation in scientific studies in the preceding year, where ionizing radiation has been used, including significant x-ray investigations.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Phenylalanine kinetics | 6 hours
  Phenylalanine balance is determined by:
  PheBal = (PheA - PheV) x F
  Where PheBal is the phenylalanine balance (mg/L), PheA is the arterial concentration of phenylalanine, PheV is the venous concentration of phenylalanine, and F is the blood flow.
Tyrosine kinetics | 6 hours
  Tyrosine balance is determined by:
  TyrBal = (TyrA - TyrV) x F
  Where TyrBal is the tyrosine balance, TyrA is the arterial concentration of tyrosine, TyrV is the venous concentration of tyrosine, and F is the blood flow.
Palmitate balance | 5 hours
  Palmitate net balance will be estimated using blood flow and arterio-venous differenves in specific activity

SECONDARY OUTCOMES:
Plasma changes in hormones and energy sources | 6 hours
  Plasma changes in the levels of insulin, glucagon, catecholamines, cortisol, IGF[1], growth hormone, glycerol, urea, glucose

CONTACTS AND LOCATIONS:
Overall Officials: Søren Laurberg, MD, DMSc, Principal Investigator — Department of Surgery P, Aarhus University Hospital
Locations (1):
- Department of Surgery P, Aarhus University Hospital, Aarhus C, Denmark